CLINICAL TRIAL: NCT04200300
Title: Professional Quality of Life in Nurses Working with Patients with Mental Disorders in Germany
Brief Title: Professional Quality of Life in German Mental Health Nursing
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Moritz Petzold, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ProQoL_P
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Mental Disorder; Burnout, Professional; Burnout, Caregiver
Keywords: Professional quality of life; Compassion satisfaction; Burnout; Nursing; Mental disorder; Mental health
MeSH Terms: conditions — Mental Disorders; Burnout, Professional; Caregiver Burden; Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nurses working with patients with mental disorders: Nurses in Germany currently working with patients with mental disorders
  Interventions: Diagnostic Test: Online questionnaire

INTERVENTIONS:
Diagnostic Test: Online questionnaire — Online questionnaire via SoSciSurvey

SUMMARY:
The purpose of this study is to assess professional quality of life in German nurses working with patients with mental disorders.

DETAILED DESCRIPTION:
The purpose of this study is to assess professional quality of life, which includes compassion satisfaction, burnout and secondary traumatization in nurses, working with patients with mental disorders, in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Nurse
* Currently working with patients with mental disorders
* At least 18 years old
* Sufficient German skills for answering the questionnaire

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses that currently work with patients with mental disorders in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Compassion Satisfaction | 1 day
  Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL) - German Version - Subscale "Compassion Satisfaction" (Minimum: 10 - Maximum: 50 - Higher scores mean a higher compassion satisfaction)
Burnout | 1 day
  Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL) - German Version - Subscale "Burnout" (Minimum: 10 - Maximum: 50 - Higher scores mean a higher level of burnout)
Secondary Traumatization | 1 day
  Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL) - German Version - Subscale "Secondary Traumatization" (Minimum: 10 - Maximum: 50 - Higher scores mean a higher level of secondary traumatization)

CONTACTS AND LOCATIONS:
Overall Officials: Moritz B Petzold, Dr., Principal Investigator — Charité Universitätsmedizin Berlin- Charité Campus Mitte - Department for Psychiatry and Psychotherapy
Locations (1):
- Charité Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapie - Charité Campus Mitte, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided